CLINICAL TRIAL: NCT03077113
Title: Pilot Study of Regional Lung Ventilation: Comparing Ventilation Images Computed From 4D CTs vs. Traditional Nuclear Medicine Ventilation Images
Brief Title: Pilot Study of Regional Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-17070
Record Dates: First submitted 2017-03-02; First posted 2017-03-10 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer; radiation therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Single Photon Emission Computed Tomography Computed Tomography; Tomography, Emission-Computed, Single-Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ventilation Images for Comparison (Other): Standard of Care: 4-D CT scan will be used to make a radiation treatment plan.
  SPECT-CT Scan: This second scan will be done on another day to make a treatment plan for comparison to the first plan.
  Interventions: Diagnostic Test: 4-D CT Scan; Diagnostic Test: SPECT-CT Scan

INTERVENTIONS:
Diagnostic Test: 4-D CT Scan — The 4-D CT scan shows how the tumor moves when patients breathe so that motion can be taken into account when planning the radiation. This is the usual way of planning lung radiation and everyone in this study will be planned using a 4-D CT scan.
  Other Names: 4-D computed tomography
Diagnostic Test: SPECT-CT Scan — It may be possible to make a more accurate plan by using a SPECT-CT scan for planning that would result in less damage to healthy lung tissue. This is not yet proven. A SPECT-CT scan uses a special camera to detect radioactivity to produce pictures which can lead to more precise information.
  Other Names: Single-photon emission computed tomography

SUMMARY:
This is a prospective study of ventilation image comparison for lung functional information incorporation in thoracic cancer treatment planning.

DETAILED DESCRIPTION:
Investigators hypothesize that a high resolution regional ventilation image (HRVI) based on 4D-CT imaging will correlate with the current low resolution state-of-the-art (SPECT-CT), which is the conventional way of measuring ventilation. HRVI may be a tool that could be widely used throughout the radiation therapy community because most radiation oncologists routinely employ 4D-CT technology in their own clinics. Investigators plan to test this hypothesis by comparing ventilation patterns on SPECT-CT images to HRVIs using a DICE analysis. As SPECT ventilation imaging is not included in our standard care, this study thus is designed as a pilot study.

Based on published data, the difference between the two methods for calculating the regional ventilation in the lower 50% ventilation volume is expected to have a standard deviation of about 0.1. Therefore, the 95% confidence interval for the difference in the regional ventilation between SPECT-CT and 4D-CT pre-treatment would have a width of no more than 0.14 if 10 patients are enrolled and as small as 0.10 when 20 patients are registered.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have early stage non-small cell lung cancer or clinical suspicion of the same in cases where the lesion is not amenable to biopsy but is enlarging and PET-positive. All patients are to be treated with stereotactic body radiation therapy as a monotherapy.
* Eligible patients must have appropriate staging studies identifying them as specific subsets of AJCC 7th edition stage I or II based on only one of the following combinations of TNM staging:

  * T1a-b, N0, M0
  * T2a, N0, M0
  * T3 (invading the chest wall, <5 cm in diameter) N0 M0
* Must be at least 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Women of childbearing potential and male participants must use an effective contraceptive method such as condom/diaphragm and spermicidal foam, intrauterine device, or prescription birth control pills.

Exclusion Criteria:

* Patients with T2b tumors or T3 tumors >5 cm or patients with tumors involving the central chest/structures of the mediastinum;
* Primary tumor of any T-stage within or touching the zone of the proximal bronchial tree, defined as a volume 2 cm in all directions around the proximal bronchial tree (carina, right and left main bronchi, right and left upper lobe bronchi, bronchus intermedius, right middle lobe bronchus, lingular bronchus, right and left lower lobe bronchi.
* Direct evidence of regional or distant metastases after appropriate staging studies
* Patients with active systemic, pulmonary, or pericardial infection;
* Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.
* Patients that receive chemotherapy (induction or sequential)
* Psychiatric or addictive disorders that impair subject's voluntary ability to participate in informed consent or protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-10-15 (Actual); Primary Completion 2015-04-16 (Actual); Study Completion 2016-08-23 (Actual)

PRIMARY OUTCOMES:
Rate of Correlation of Ventilation Images | Up to 1 year
  The primary objective is to compare the regional ventilation using SPECT-CT and that as determined from the pre-treatment 4D-CT routinely collected at simulation in lung/abdominal patients (standard of care). 50% of the lower portion lung image will be used for the purpose of determining the regional ventilation for this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dilling, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/